CLINICAL TRIAL: NCT02030340
Title: In Vivo Comparison of Air Charged Catheters With Water Filled Catheters for Intravesical and Intrarectal Pressures Recording During Urodynamic Study
Brief Title: Comparison of Air Charged Catheters With Water Filled Catheters for Urodynamic Study
Acronym: ACWF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: UMCUtrecht, department of Urology (Unknown); T-Doc-LLC (Unknown)
Responsible Party: Principal Investigator, Peter F.W.M. Rosier, Senior Lecturer MD PhD, UMC Utrecht
Other Study IDs: AC-WF; T-Doc-LLC (Other Grant/Funding Number: T-Doc-LLC Wilmington USA)
Record Dates: First submitted 2013-03-06; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Incontinence
Keywords: urodynamic investigation; lower urinary tract dysfunction; catheter; air-charged; water filled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Testing Lower urinary tract dysfunction: All patients with lower urinary tract dysfunction where urodynamic diagnosis is required according to standards and (international) practice guidelines will have a synchronous double system (combination of air-charged and water filled) urodynamic test.
  Interventions: Procedure: lower urinary tract dysfunction

INTERVENTIONS:
Procedure: lower urinary tract dysfunction — Urodynamic investigation with a double (two systems: air-charged and water filled) catheter system
  Other Names: T-doc air charged catheters.

SUMMARY:
Various systems to measure intravesical and intrarectal pressure during urodynamic testing; especially cystometry, exist. Water filled tube -systems are the most commonly used and should be regarded as the contemporary standard. A water filled system is however sensitive to tube and or patient movement artefacts and prone to erroneous calibration. Air charged catheters are less sensitive to patient and especially tubing- movements, and calibrate easier. However, in vitro tests have demonstrated that air charged catheters respond somewhat slower and relatively damped, especially to rapid pressure changes as in (simulated) coughing, in comparison with water filled systems. The clinical relevance of these observations is unknown.

This is a study to compare the technical reliability and clinical applicability of the two types of catheter systems for cystometry in a synchronous double catheter testing procedure in a prospective group or patients scheduled for urodynamic investigation.

DETAILED DESCRIPTION:
Study design: Patient cohort, acute experiment, mono -center synchronous double urodynamic catheter technique study.

Study population: Adult female patients and male or female patients with spinal cord injury or meningomyelocele unable to void, scheduled for urodynamic investigation on the basis of contemporary standards and guidelines, because of signs and or symptoms of lower urinary tract dysfunction.

Intervention: Synchronous double catheter urodynamic testing; Standard filling cystometry with both air-charged ánd water filled catheter pairwise inserted, and connected to the registry equipment.

Main study parameters/endpoints: Difference of intravesical pressure increment maximum during filling cystometry between the two systems.

Primary hypothesis to test: The average difference as well as the average absolute difference of maximum water pressure (standard system) and maximum air pressure (comparator) are both 0 (zero).

There is no per-protocol for follow up of the patients.

ELIGIBILITY:
Inclusion Criteria:

(All necessary:)

* Female gt18 years
* Scheduled for urodynamic investigation on the basis of contemporary standards and guidelines, because of signs and symptoms of lower urinary tract dysfunction.
* May perform (not excluded) intermittent (self) catheterisation.
* No signs of voiding dysfunction (routine outpatient max flow above 20 millilitre per second without postvoid residual)
* No signs of bladder /pelvic pain syndrome

OR:

(All necessary)

* Male or female gt18years
* Complete spinal cord injury, level above T12, or meningomyelocele unable to void and significantly reduced or no pelvic floor, urethral or bladder sensation.
* May have (not excluded) 'sacral sparing'; some residual anal sensation
* Scheduled for urodynamic investigation on the basis of contemporary standards and guidelines, because of signs and symptoms of lower urinary tract dysfunction or because of routine (protocol, guidelines) follow -up.
* Usually: performing intermittent (self) catheterisation); not excluded.
* May have (not excluded) indwelling catheter.

Exclusion Criteria:

* Unwilling or unfit to sign informed consent.
* American Society of Anesthesiologists -score gt2; karnovsky lt80percent.
* Male with normal lower urinary tract sensation.
* Women with signs of voiding dysfunction.
* Patients included in scientific studies (for other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled (on the basis of contemporary clinical standards and protocols) for standard urodynamic investigation.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The difference between the water filled catheter recorded and simultaneously air charged catheter recorded maximum pressure (amplitude)during the bladder filling phase of urodynamic test. | acute comparison during one test with two types of catheter
  Null hypothesis: the (absolute mean) difference between the water filled catheter recorded and simultaneously air charged catheter recorded maximum pressure (amplitude) observed with a dominant detrusor pressure event during urodynamic filling as obtained with both systems is close to zero.

SECONDARY OUTCOMES:
responses to relevant pressure events: end fill pressure, maximum contraction pressure, maximum pressure at overactive detrusor contraction and maximum cough pressure. | acute comparison during one test with two types of catheter
  to test the clinical feasibility (-mean absolute- pressure responses differences) of the air charged system, against the contemporary clinical standard. Perfect feasibility of air charged catheter system is achieved when the measured pressures are equal (difference zero) to the water filled system in all performed measurements in all situations.

CONTACTS AND LOCATIONS:
Overall Officials: Peter FW Rosier, MD PhD, Principal Investigator — University Medical Center Utrecht, the Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Rosier PF, Gajewski JB, Sand PK, Szabo L, Capewell A, Hosker GL; International Consultation on Incontinence 2008 Committee on Dynamic Testing. Executive summary: The International Consultation on Incontinence 2008--Committee on: "Dynamic Testing"; for urinary incontinence and for fecal incontinence. Part 1: Innovations in urodynamic techniques and urodynamic testing for signs and symptoms of urinary incontinence in female patients. Neurourol Urodyn. 2010;29(1):140-5. doi: 10.1002/nau.20764. PMID 19693949